CLINICAL TRIAL: NCT06052969
Title: PERFUSION AIS - Pulse Endovascular ReperFUSION for Acute Ischemic Stroke: An Early Feasibility Clinical Study
Brief Title: Pulse Endovascular ReperFUSION for Acute Ischemic Stroke
Acronym: PERFUSION AIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Euphrates Vascular, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MED-CLN-001P; G220131/S001 (Other: U.S. Food and Drug Administration Center for Devices and Radiological Health)
Record Dates: First submitted 2023-09-11; First posted 2023-09-25 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Acute Ischemic Stroke AIS; Cerebral Arterial Disease
Keywords: MicroBeads; Pulse NanoMed System
MeSH Terms: conditions — Cerebral Arterial Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, single-arm early feasibility study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Group/Cohort (Experimental): Subjects presenting to the emergency department with AIS, eligible for thrombolytic therapy, and with evidence of an occlusive clot by angiographic imaging will be considered for inclusion in the study. Post-thrombolytic therapy and mechanical thrombectomy eligible Subjects will receive the experimental NanoMED device.
  Interventions: Device: Pulse NanoMED System

INTERVENTIONS:
Device: Pulse NanoMED System — The Pulse NanoMED System is comprised of iron nanoparticles and a small, portable, magnetic Workstation.

SUMMARY:
Prospective, multi-center, single-arm early feasibility study enrolling a minimum of 15 subjects at up to a minimum of 3 active investigational sites in the United States.

The subjects must be diagnosed with acute ischemic stroke (AIS), must be post-mechanical thrombectomy, will have had intravenous thrombolytics, and have a visible MCA, ACA or PCA occlusive clot on initial angiographic imaging.

Each subject will receive the Pulse NanoMED procedure after attempted neurovascular therapy to achieve better reperfusion.

ELIGIBILITY:
Inclusion Criteria:

1. The participant provides written informed consent using an Informed Consent Form (ICF) that is reviewed and approved by the Institutional Review Board (IRB) or an acceptable patient surrogate.
2. The participant is ≥ 18 years old and less than 85 years old.
3. Patients with symptomatic large vessel occlusion (LVO) who undergo MT as part of their standard of care and have residual occlusion involving the anterior, middle or posterior cerebral arteries resulting in a eTICI score greater than 2b50 at the end of the procedure with three or less MT device passes.
4. Estimated delay to onset of rescue Pulse NanoMED MicroBead administration <9 hours from symptom onset, defined as the point in time the patient was last known well (LKW).
5. Post-MT and has had thrombolytic therapy <9 hours prior to the proposed start time of System therapy
6. No significant pre-stroke functional disability (modified Rankin scale 0-1)
7. Baseline NIHSS≥6
8. ASPECTS >6 on non-contrast CT (NCCT) scan if symptoms lasting <8 hours
9. CT-Perfusion (CTP) is optional, if performed, should demonstrate rCBF <30% lesion volume ≤70 mL.
10. Imaging should be obtained within 75 minutes of the onset of mechanical thrombectomy.

Exclusion Criteria:

1. NIHSS score on admission >25
2. Use of carotid artery stents during the endovascular procedure requiring dual antiplatelet therapy
3. Female who is pregnant or lactating or has a positive pregnancy test at the time of admission
4. Current participation in another investigational drug or device treatment study
5. Known allergy or sensitivity to iron
6. Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency
7. Known coagulopathy, INR >1.7, or use of novel anticoagulants <12h from symptom onset
8. Known Platelets <100,000
9. Known Renal Failure as defined by a serum creatinine >3.0 mg/dl (or 265.2 μmol/l) or glomerular Filtration Rate [GFR] <30
10. Subject who requires hemodialysis or peritoneal dialysis or who has a contraindication to angiogram for whatever reason
11. Any hemorrhage on CT/MRI
12. Clinical presentation suggests a subarachnoid hemorrhage, even if initial CT or MRI scan is normal.
13. Suspicion of aortic dissection
14. Subject currently uses or has a recent history of illicit drug(s) or abuses alcohol.
15. History of life-threatening allergy (more than rash) to contrast medium
16. SBP >185mmHg or DBP >110mmHg refractory to treatment
17. Serious, advanced, terminal illness with anticipated life expectancy <6 months
18. Pre-existing neurological or psychiatric disease that would confound evaluation
19. Presumed vasculitis or septic embolization
20. Known sensitivity or allergy to contrast materials that cannot be previously treated properly
21. The subject takes Coumadin and its interruption could compromise their safety
22. Known allergy or contraindication to double antiplatelet treatment
23. Known hypersensitivity or contraindication to iron or polyethylene glycol-based agents
24. Known contraindication to MRI (examples include, but are not known, implantable cardioverter-defibrillator, pacemaker, clip-on or spiral aneurysm, neurostimulator)
25. The physical geometry of the subject that prevents the placement of the magnet
26. The subject has signs or symptoms of systemic infection/sepsis (temperature of ≥38.0 Celsius and/or white blood cell count of ≥12,000 cells/uL). If the subject has a localized infection, such as cellulitis or osteomyelitis, or the infection is properly treated and controlled, according to the discretion of the researcher, the patient can enroll
27. Known or suspected cardiovascular condition that causes a secondary or tertiary heart block, tachycardia-bradycardia syndrome, or symptomatic postural hypotension requiring medical intervention
28. Known or suspected symptomatic hemochromatosis or hemosiderosis
29. Known or suspected liver disease, such as hepatitis and/or cirrhosis
30. The subject has received iron replacement therapy or contrast for iron-based MRI in the previous 30 days

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 24 hours, 7 days (or discharge, if earlier), 30 days, and 90 days post-procedure
  To test the safety and feasibility of the Pulse NanoMED System in ischemic stroke patients. The potential clinical benefit of early recanalization will be visually assessed by a core laboratory by comparing baseline DSA, CTA, or MRA images with images taken at set timepoints.

SECONDARY OUTCOMES:
Secondary Objective | 24 hours, 7 days (or discharge, if earlier), 30 days, and 90 days post-procedure
  To test the hypothesis that ischemic stroke patients that receive thrombolytic therapy and endovascular therapy will have improved reperfusion as assessed by eTICI and clinical outcomes when provided adjunctive treatment with the Pulse NanoMED System.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina - Prisma, Columbia, South Carolina, United States